CLINICAL TRIAL: NCT01394263
Title: Phase III, Open-Label Randomized, Parallel, Active-Control Study to Evaluate Efficacy and Safety of Histrelin Subdermal Implant in Patients With Metastatic Prostate Cancer
Brief Title: Study of Histrelin Subdermal Implant in Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 302
Record Dates: First submitted 2011-07-13; First posted 2011-07-14 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer; Adenocarcinoma of the Prostate
Keywords: prostate cancer; PSA; testosterone suppression
MeSH Terms: conditions — Prostatic Neoplasms | interventions — histrelin; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zoladex goserelin implant. (Active Comparator): Zoladex goserelin implant: D, L-lactic and glycolic acids copolymer. Injected subcutaneously into the upper abdominal wall.
  Interventions: Drug: Zoladex goserelin implant
- Histrelin Acetate implant (Experimental): Histrelin hydrogel implant, 3 cm x 3.5 mm, containing 50 mg of histrelin acetate, surgically placed subdermally into the inner aspect of the upper arm.
  Interventions: Drug: Histrelin hydrogel implant

INTERVENTIONS:
Drug: Histrelin hydrogel implant — 50 mg histrelin acetate in hyrogel implant
  Other Names: Vantas
  Arms: Histrelin Acetate implant
Drug: Zoladex goserelin implant — goserelin implant injection.
  Other Names: Zoladex
  Arms: Zoladex goserelin implant.

SUMMARY:
This trial was an open-label, multi-national, randomized, parallel treatment, active-control multicenter study in adult males with documented metastatic prostate cancer disease who were judged to be candidates for hormone therapy.

DETAILED DESCRIPTION:
This trial was an open-label, randomized, parallel treatment, active-control multicenter study in adult males with documented metastatic prostate cancer disease who were judged to be candidates for hormone therapy.

Within 21 days prior to implant insertion, all prospective enrollees were entered into a screening period to provide medical history, demographic information, physical examination, laboratory evaluations, 12-lead ECG, bone scan, chest x-ray, liver ultrasound, concomitant medications and procedures, and a physician assessment including pain level and WHO performance scale in order to assess eligibility for the study. Written informed consent was obtained before any procedures were undertaken.

Once inclusion/exclusion criteria were met, baseline evaluations (physical assessment and examination, vital signs and weight, clinical laboratory evaluations, concomitant medications and procedures, adverse events, and a Quality of Life questionnaire) were obtained prior to implant insertion on Day 1 [Visit 1]. All appropriately screened patients were to then receive either histrelin acetate 50-mg or Zoladex 3-Month 10.8 mg implant based on 1:1 randomization at Day 1 [Visit 1]. Patients with implants were evaluated at Week 1 and 2 [Visits 2 and 3] post-insertion for testosterone and PSA concentrations, vital signs, adverse events, and concomitant medications and procedures. The Zoladex implants were replaced at Weeks 12, 24, 36, and 48 [Visits 6, 9, 12, and 15], while the histrelin acetate implants were replaced at Week 52 (Visit 16), respectively. Patients were followed monthly from Weeks 4 to 60 [Visits 4 to 18] to evaluate testosterone and PSA concentrations, adverse events, concomitant medications and procedures, disease progression, and urine and serum histrelin in the renal/hepatic impairment subgroup. Periodic clinical and subjective assessments were completed for all patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Male patients with histologically confirmed adenocarcinoma of the prostate
* Disease staging of M1 or apparent failure of the initial definitive therapy (e.g., prostatectomy, radiation, etc.), suggested by either an elevated PSA (5 ng/mL or greater within the previous 28 days), or when below 5ng/mL, rising PSA values (elevation from previous measurement greater than or equal to 0.1 ng/mL on three consecutive measurements at least two weeks apart with at least one of these measurements being within the last 28 days which may include the Screening Visit result, if needed)
* Clinically indicated for androgen suppression therapy
* Age 45 years or older
* Serum testosterone level of 150 ng/dL (5.25 nmol/L) or greater at screening
* PSA level of 5ng/mL or greater within the previous 28 days, or an increase in PSA (elevation from previous measurements greater than or equal to 0.1ng/mL on three consecutive measurements at least two weeks apart)

Key Exclusion Criteria:

* Bilateral orchiectomy
* Prior androgen-ablative or systemic corticosteroid therapy within the past year
* Second malignancy within five years, except adequately treated nonmelanomatous skin cancer or superficial bladder cancer
* Spinal cord compression
* Location of vertebral metastases that indicate risk of spinal cord compression during initial treatment period in the opinion of the Investigator
* Brain metastasis previously confirmed by CT scan

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2000-05; Primary Completion 2001-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Suppression of testosterone via the percent of patients whose testosterone was at or below chemical castration levels (<=50 n/dL) through 52 weeks of treatment. | 52 weeks

SECONDARY OUTCOMES:
Secondary efficacy was assessed by serum LH, PSA, and PAP, WHO Performance Status, Pain Level assessment, the National Prostatic Cancer Project (NPCP) assessment for objective clinical status, PSA status, time to disease progression, and QoL. | 52 weeks